CLINICAL TRIAL: NCT03569644
Title: Creation of a Tool to Assess Quality of Life in Patient With Auto-inflammatory Diseases
Brief Title: Quality of Life in Patients With Auto-inflammatory Diseases
Acronym: MAI-PATIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K160903J; 2017-A02673-50 (Other: ANSM)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Autoinflammatory Diseases
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases

STUDY DESIGN:
Intervention Model Description: The study is based on interviews that will be recorded in digital audio and then transcribed literally. The consultation for this research is 45 to 90 minutes long. This prolongs their presence in consultation with the doctor. For this reason, the study was classified as Interventional according to French regulations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- qualitative study (Other): heterogeneous group of patients
  Interventions: Other: qualitative study

INTERVENTIONS:
Other: qualitative study — Interviews

SUMMARY:
This qualitative interview-based study aim to build a tool to assess quality of life in patients (adults or children) suffering from 6 autoinflammatory diseases (FMF, TRAPS, CAPS, MKD, Still and PFAPA).

DETAILED DESCRIPTION:
Recent understanding of the physiopathological mechanisms that underpin autoinflammatory diseases (AIDs) allowed a revolution in the therapeutic management of these patients, particularly through the use of biotherapies. However new treatments need to be evaluated by valid tools. AIDAI score created and validated by our team evaluates activity of 4 autoinflammatory diseases. One of the important components, not explored by the scores currently available, is the impact of these treatments on quality of life (QoL) of patients. The existing quality of life scales are not adapted to these recurrent chronic pathologies. Throught a qualitative study based on interviews of patients and/ or parents, the investigators aim to build a tool to evaluate QoL in patients suffering from 6 aAIDs :familial Mediterranean fever (FMF), mevalonate kinase deficiency (MKD), tumour necrosis factor receptor-associated periodic syndrome (TRAPS), cryopyrin-associated periodic syndromes (CAPS), Still's disease and PFAPA syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Any patient (child and adult) with one of the 6 AIDs (FMF, TRAPS, MKD or CAPS, PFAPA or Still's disease) regardless of the activity of the disease. The diagnosis will have been made by the referring physician according to criteria specific to each AIDs
* Volunteer to participate in the study
* With at least one parent present at the consultation if it is a child under 18 years old
* For minors, agreement of the parents or their legal representative or one of the present parents
* Information for children as far as their age and condition allow
* Affiliation to a national health insurance.

Exclusion Criteria:

* patient or relative (according to age)refuse to participate.
* Bad understanding of French.
* Other chronic inflammatory pathology associated (example: Crohn's, SPA, uveitis, psoriasis ...)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Qualitative evaluation of quality of life by interviews of patients and/or parents | 45 to 90 min
  The interviews will be recorded in digital audio and then transcribed literally. The analysis will be phenomenological. Four age group will be interviewed : < 6 year-old (parents), 6 to 12 year-old (patients and parents) , 13 to 17 year-old (patients and parents) , > 18 year-old (patients)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH André Mignot, Le Chesnay, France
  - TENON, Paris, Paris
  - Dr Maryam PIRAM, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: Undecided